CLINICAL TRIAL: NCT03649425
Title: COMPARATIVE PROSPECTIVE STUDY OF SURFACE AND DEEP COMPLICATIONS FOUND IN THE PINS OF EXTERNAL FIXERS COMPARING STEEL PINS AND PINS COATED WITH HYDROXIAPATITA
Brief Title: COMPARATIVE PROSPECTIVE STUDY OF COMPLICATIONS FOUND IN THE PINS OF EXTERNAL FIXERS COMPARING STEEL PINS AND PINS COATED WITH HYDROXIAPATITA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Collaborators: Instituto de Ortopedia e Traumatologia de Passo Fundo (Unknown); Universidade de Passo Fundo (Other)
Responsible Party: Sponsor
Other Study IDs: 84939418.6.0000.5342
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-05

CONDITIONS: External Fixation Pin Site Infection
Keywords: infection; pin site; external fixator; hydroxyapatite coated
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- hydroxyapatite coated pins: Patients submitted to surgical treatment with external fixators using pins coated with hydroxyapatite.
- uncoated steel pins: Patients submitted to surgical treatment with external fixators using uncoated steel pins.

SUMMARY:
The present study is a prospective non-randomized and comparative study of patients undergoing surgical treatment with external fixators of any type, between May 2018 and May 2020, in the city of Passo Fundo, RS, Brazil, in the São Vicente de Paulo hospitals. A study in which we compared infection rates, pin loosening and complications found in external fixators made with hydroxyapatite coated pins and uncoated steel pins.

DETAILED DESCRIPTION:
We will use as a guide to define the degree of infection and the conduct to be taken in the classification of Mas Oxford Nuffield (Table 3), therefore the presence of infection occurring in patients classified as Grade 2 - erythema of the skin, serous or purulent secretion, pain and sensitivity in soft tissues capable of mobilizing with analgesia. We will also send to the culture the tip of two pins removed from each patient to evaluate possible colonization and to compare with the degree of classification presented in the pin in question, we will do this with a pin without signal of infection and with the pin with the highest degree of classification presented in each patient at the time of the external fixator removal.

We will use as a method of insertion of the pin the pre-perforation irrigated before the insertion of the pins, to decrease the chances of thermal necrosis and consequent release or infection. We will use steel Shanz pins coated with hydroxyapatite or not in size between 5-6mm. Comorbidities and risk factors such as diabetes mellitus, smoking, immunodepression, among others, will be computed for later comparison with the data collected. The degree of classification of the fractures, as well as the pathologies that were treated with the fixators, as well as the residence time with the external fixator will also be computed for later comparison with the data collected.

For the elaboration of this study, the patients will be prospectively observed, which will be submitted to the treatment of several pathologies with external fixators, of any type. The occurrence of infection and / or loosening of the pins, as well as the influence of risk factors and the cultural examination results of the pins removed at the end of the treatment will be recorded. The objectives of the study are to comparatively evaluate the differences in complications of infection, pin loosening and microbiological results of cultural examinations, between patients submitted to external fixators with uncoated steel pins and steel pins coated with hydroxyapatite. The influence of risk factors on outcomes will also be observed.

ELIGIBILITY:
Inclusion Criteria:

* We will select for the study patients who agree to participate, signing the commitment term for data use, and who underwent surgical treatment with external fixation of any type both for fracture treatment and correction of deformities, treatment of osteomyelitis and or pseudoarthrosis , for a minimum period of 2 weeks.

Exclusion Criteria:

* We will exclude patients who do not agree to participate in the study, patients who have had external fixation for less than 2 weeks, and patients in whom we have lost follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent surgical treatment with external fixators for at least 2 weeks, regardless of age, gender and comorbidities.
Sampling Method: Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-11-25 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
compare infectious complications | April 2018 and December 2019
  To compare superficial and deep infectious complications associated with the presence of external fixation pins. To evaluate the incidence and degree of infection at pin insertion sites, osteomyelitis and wound infection, comparatively between hydroxyapatite and uncoated pins.
Evaluate the incidence of loosening of the pins | April 2018 and December 2019
  To evaluate the incidence of pin loosening, comparatively between pins coated with hydroxyapatite and uncoated pins, in the external fixators.

SECONDARY OUTCOMES:
risk factors and comorbities associated | April 2018 and December 2019
  To evaluate the risk factors and comorbidities associated with infectious complications and pin loosening in the patients participating in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided